CLINICAL TRIAL: NCT02419846
Title: The Effectiveness of a Proposed Prostate Cancer Outreach Program in a Predominantly African American Community That Promotes Informed Decision-making for Prostate Cancer Screening and Utilizes Community Navigation
Brief Title: Informed Decision Making Intervention in Screening for Prostate Cancer of Predominantly African American Participants in a Community Outreach Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit due to COVID limitations / Funding Unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CASE3815
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Prostate Carcinoma
Keywords: Informed Decision Making; Prostate; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Early Intervention, Educational; Methods; Program Evaluation; Prostate-Specific Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men over 40: Screening with intervention (Experimental): Participants over the age of 40 complete an educational intervention comprising a 10-20 minute PowerPoint presentation given by an experienced healthcare professional that discusses prostate cancer facts, screening guidelines, risks, benefits, and consequences. Participants may undergo a screening exam comprising a prostate specific antigen level and digital rectal exam.
  Interventions: Other: Educational Intervention; Procedure: digital rectal examination; Other: Pre-test administration; Other: Survey Administration; Other: Prostate-specific antigen measurement; Other: Post test administration
- Men 18-39: Educational intervention (Experimental): Participants between 18 and 39 complete an educational intervention comprising a 10-20 minute PowerPoint presentation given by an experienced healthcare professional that discusses prostate cancer facts, screening guidelines, risks, benefits, and consequences.
  Interventions: Other: Educational Intervention; Other: Pre-test administration; Other: Survey Administration; Other: Post test administration

INTERVENTIONS:
Other: Educational Intervention — Attend 10-20 minute PowerPoint presentation that will discuss prostate cancer facts, screening guidelines, risks, benefits, and consequences
  Other Names: PowerPoint Presentation; Intervention, Educational
Procedure: digital rectal examination — Undergo digital rectal exam by a licensed healthcare professional. The results of this exam will be subjective as per clinician; however, will be coded as normal or abnormal. This is considered standard of care for prostate cancer screening
  Other Names: DRE
  Arms: Men over 40: Screening with intervention
Other: Pre-test administration — 15 questions which test participants' knowledge of prostate cancer according to ACS guidelines. Questions will be multiple choices and true/false/unsure answers
  Other Names: questionnaire administration
Other: Survey Administration — Survey will be administered at the end of the program for participants to assess their experience
  Other Names: Program Evaluation
Other: Prostate-specific antigen measurement — PSA levels will be drawn and run as per institutional Laboratory standards. Criteria for referral and follow up will be assessed as per National Comprehensive Cancer Network (NCCN) guidelines
  Other Names: PSA levels
  Arms: Men over 40: Screening with intervention
Other: Post test administration — Post test will include the same 15 questions as on the pretest to assess for improvement in knowledge and understanding
  Other Names: questionnaire administration

SUMMARY:
This clinical trial studies an informed decision making intervention of screening for prostate cancer in predominantly African American participants. It also evaluates participants' knowledge about prostate cancer screening and to improve understanding. Using decision aids such as culturally sensitive written material, verbal information, and videos to educate patients about screening may increase patient participation and knowledge. This may increase confidence in participants' decisions. Raising awareness about prostate cancer in the communities may increase the participants' willingness to be screened for prostate cancer once they have learned about it.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

(A) To assess the effectiveness of a proposed educational model for informed decision about Prostate Cancer in high risk men over age 40 which compares informed decision making and shared decision making (B) to improve knowledge about prostate cancer in men over age 18

OUTLINE:

Participants complete an educational intervention comprising a 10-20 minute PowerPoint presentation given by an experienced healthcare professional that discusses prostate cancer facts, screening guidelines, risks, benefits, and consequences. Some participants then undergo a screening exam comprising a prostate specific antigen level and digital rectal exam.

After completion of study, participants are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of 18 will be asked to participate in the educational component of the program; men over the age of 40 will be offered the screening component after the educational portion of the event; participants over age of 40 will have the opportunity to make an informed decision in regards to prostate cancer screening based on this information and the educational material; American Cancer Society (ACS) guidelines recommend having a discussion about screening in men who have an expected mortality of greater than 10 years; data on comorbidities and 10-year mortalities will be collected on every participant using the University of California at San Francisco (UCSF) mortality index
* Educational component: men over the age of 18
* Screening component: men over age 40

Exclusion Criteria:

* Known personal history of prostate cancer
* Active malignancy, metastatic disease, or anyone undergoing treatment for malignancy

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants over age 18 that demonstrate improved knowledge about prostate cancer screening | Up to 1 year
  Improved understanding will be defined as an increase in the number of correct answers seen on the post Prostate Screening Education Questionnaire. The underlying likelihood of a positive response, or improved understanding of prostate cancer screening, can be estimated using a 95% confidence interval that has a maximum half-width of 6%.
Proportion of participants over age 40 who find this education and screening model helpful in making an informed decision about prostate cancer screening as measured by the satisfaction survey questions | Up to 1 year
  Helpfulness of the program will be measured on a 5-point Likert scale where the two uppermost categories are considered a positive response.

SECONDARY OUTCOMES:
Proportion of participants who choose to enter the clinical trial | Up to 1 year
Proportion of participants who choose screening after educational intervention | Up to 1 year
10-year expected mortality based on USCF 10-year Mortality Index for all participants | Up to 1 year
Proportion of participants with a high 10-year mortality based on UCSF index who choose to be screened for prostate cancer after educational intervention | Up to 1 year
Proportion of abnormal results found with screening and referred to follow-up assessed as per National Comprehensive Cancer Network guidelines | Up to 1 year
Proportion of participants diagnosed with malignancy based on follow up biopsies and work-up during the course of the study | Up to 1 year
Proportion of participants with family history of prostate cancer | Up to 1 year
Proportion of participants referred to a primary care physician who did not previously have a primary care physician | Up to 1 year
Proportion of participants who asked the physician to make a decision for them in spite of educational intervention | Up to 1 year
Proportion of participants who expressed satisfied with this proposed informed consent and education model | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Samir Abraksia, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States